CLINICAL TRIAL: NCT05842278
Title: The Dosage Effect of Personalized Brain Functional Sectors(pBFS) Guided rTMS Treatment for Major Depressive Disorder： a Randomized， Double-Blind， Sham-controlled Trial
Brief Title: The Dosage Effect of pBFS Guided rTMS Treatment for MDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Collaborators: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLMDDhlg1
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Moderate Depression; Major Depressive Disorder; Severe Depression
Keywords: transcranial magnetic stimulation, rTMS; Major Depression, Moderate Depression, MDD; personalized neuromodulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 4 session rTMS (Active Comparator): Four sessions of active rTMS would be delivered to the left DLPFC daily, with a session of 1800 pulse.
  Interventions: Device: 4 session rTMS
- 6 session rTMS (Active Comparator): Six sessions of active TMS would be delivered to the left DLPFC daily, with a session of 1800 pulse.
  Interventions: Device: 6 session rTMS
- 8 session rTMS (Active Comparator): Eight sessions of active rTMS would be delivered to the left DLPFC daily, with a session of 1800 pulse.
  Interventions: Device: 8 session rTMS
- 10 session rTMS (Active Comparator): Ten sessions of active rTMS would be delivered to the left DLPFC daily, with a session of 1800 pulse.
  Interventions: Device: 10 session rTMS
- sham rTMS (Sham Comparator): Subjects were randomized to receive 4 sessions or 6 sessions or 8 sessions or 10 sessions of sham rTMS to the left DLPFC daily in a 1:1:1:1 ratio.
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: 4 session rTMS — Participants will receive 4 sessions per day of 1800 pulses per session, lasting for 5 days. Individualized targets will be generated using the pBFS method.
  Arms: 4 session rTMS
Device: 6 session rTMS — Participants will receive 6 sessions per day of 1800 pulses per session, lasting for 5 days. Individualized targets will be generated using the pBFS method.
  Arms: 6 session rTMS
Device: 8 session rTMS — Participants will receive 8 sessions per day of 1800 pulses per session, lasting for 5 days. Individualized targets will be generated using the pBFS method.
  Arms: 8 session rTMS
Device: 10 session rTMS — Participants will receive 10 sessions per day of 1800 pulses per session, lasting for 5 days. Individualized targets will be generated using the pBFS method.
  Arms: 10 session rTMS
Device: sham rTMS — The parameters in the sham arms are the same as the active stimulation groups. Stimulation was delivered by the same device as the active group fitted with a sham coil.
  Arms: sham rTMS

SUMMARY:
The investigators aim to find the optimal dosage of the pBFS-guided rTMS treatment for patients with moderate to severe depression.

DETAILED DESCRIPTION:
In 2022, the FDA cleared a large dosage of repetitive transcranial magnetic stimulation for treatment-resistant depression (TRD), which requires 10 sessions per day of 1,800 pulses per session for a total of 18,000 pulses per day. The inter-session interval is 50 min, and it costs patients 9 hours for the intervention. The investigators assume that patients with moderate to severe depression may not need 10 sessions per day, patients may achieve response or remission with a less amount of dosage, which will save the cost of treatment. Hence, the investigators try to find the optimal treatment dosage for patients with moderate to severe depression.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner in a 1:1:1:1:1 ratio to each active rTMS group with different pulses (4×1800 pulses, 6×1800 pulses, 8×1800 pulses, 10×1800 pulses) and sham-control group. And then all participants will undergo a 5-day rTMS treatment followed by four- and eight weeks follow-up visits. Participants will keep a stable treatment regime during treatment and the four-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized/outpatient patients aged 18-65 years (inclusive), male or female.
* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for depression disorder without psychotic symptoms, and currently experiencing a recurrence episode.
* Total HAMD17 score ≥20 before randomization.
* Total MADRS score of ≥25 before randomization.
* Inadequate response to at least one antidepressant trial of adequate doses and duration.
* Participants currently are on a stable or no-drug use for at least 4 weeks before randomization. The type and dose of antidepressant drugs remained unchanged throughout the intervention period.
* Voluntarily participate in the trial and able to provide informed consent. Able to comply with the planned visit, examination and treatment plan, and other study procedures.

Exclusion Criteria:

* Meet DSM-5 diagnostic criteria for other mental disorders (such as schizophrenia spectrum disorders, bipolar and related disorders, neurodevelopmental disorders, neurocognitive disorders, or depressive disorders due to substances and/or medications, depressive disorders due to other medical problems, etc.);
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* Patients with serious or unstable diseases of the cardiovascular, liver, kidney, blood, endocrine, neurological system, and other systems or organs, especially those with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, VNS, DBS, tDCS, light therapy, or other physical therapy related to mental illness within 3 months;
* Currently receiving or plan to start formal cognitive or behavioral therapy, or systemic psychological therapy (interpersonal therapy, dynamic therapy, cognitive behavioral therapy, etc.) during the trial;
* Substance abuse or dependence (including alcohol, drugs, and other psychoactive substances) in the past 1 year;
* Female of childbearing potential who plans to become pregnant during the trial.
* Female that is pregnant or breastfeeding.
* Patients in any clinical trials of other drugs or physical therapy within 1 month before the screening.
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from baseline to Immediate Post-treatment | Baseline, Day 5(Immediate Post-treatment)
  The MADRS is a validated instrument stratifying the severity of depressive episodes in adults. The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression).

SECONDARY OUTCOMES:
Change in MADRS | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment, 56 days Post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression.
Change in Hamilton Depression Scale (HAMD-17) | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment, 56 days Post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The Hamilton Depression Rating Scale (HDRS, or Ham-D) is the most widely used clinician-administered depression assessment scale. The Ham-17 version consists of 17 items assessing mood, guilt, general somatic symptoms, work and activities, anxiety, and slowness of thought and speech. Each item is scored on a scale of 0 to 4, except for the somatic, sleep, and insight items which are scored 0 to 2. On the HAM-17 there can be a total score of 22. Higher scores represent higher depression severity.
Change in Quick Inventory of Depressive Symptomatology Self-Report (QIDS_SR) | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment, 56 days Post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The 16-item QIDS_SR is a widely used self-report instrument covering depressive symptoms incorporating nine Diagnostic and Statistical Manual of Mental Disorder-IV (DSM-IV) diagnostic criteria for major depressive disorders. Each item is scored on a scale of 0 to 4. Higher scores represent higher depression severity.
Safety estimated using SSI, YMRS | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment, 56 days Post-treatment
  Scale for Suicide Ideation (SSI) measures suicide ideation, Young Mania Rating Scale(YMARS) measures mania

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality, China